CLINICAL TRIAL: NCT05670067
Title: Localized Alveolar Ridge Reconstruction and Soft Tissue Augmentation Using a Triple Graft From the Maxillary Tuberosity Simultaneous With Immediate Implant Placement ( a Randomized Clinical Clinical Study)
Brief Title: Alveolar Ridge and Soft Tissue Augmentation Using Graft From the Maxillary Tuberosity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Hesham Mohamed, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: no 948
Record Dates: First submitted 2022-12-11; First posted 2023-01-04 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Immediate Implant Placement
MeSH Terms: interventions — Transplantation, Autologous; Bone Transplantation; Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: two group in which the same procedure is done ( immediate implant placement) using different bone grafts
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor will not know the grouping of the study he will only know that immediate implant was placed in both groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant with bone graft (autogenous) (Active Comparator): with immediate implant placement autogenous grafting using maxillary tuberosity will be done
  Interventions: Procedure: maxillary tuberosity bone graft (autogenous graft)
- immediate implant with bonegraft (xenograft) (Active Comparator): with immediate implant placement grafting with xenograft will be done
  Interventions: Procedure: Bone graft (xenograft)

INTERVENTIONS:
Procedure: maxillary tuberosity bone graft (autogenous graft) — the usage of maxillary tuberosity as source of autogenous graft supplying the needed cells for bone regeneration
  Arms: immediate implant with bone graft (autogenous)
Procedure: Bone graft (xenograft) — xenograft is bone graft material that is obtained from porcine, bovine or equine source
  Arms: immediate implant with bonegraft (xenograft)

SUMMARY:
In the study immediate implant is placed in the anterior region with autogenous bone grafting from the maxillary tuberosity in one group and in the other group immediate implant is placed with xenograft .IN both groups soft tissue grafting is done using connective tissue assessment of buccal bone thickness and soft tissue will be done 6 months post operative

DETAILED DESCRIPTION:
immediate implant will be placed in the anterior region with autogenous graft from the maxillary tuberosity and in the other group immediate implant will be laced with xenograft soft tissue grafting using sub-epithelial connective tissue will in both groups assessment of buccal bone thickness is the primary outcome of the study, while volumetric assessment of the soft tissue and patient satisfaction are the secondary and tertiary outcome the assessment of all outcome will be 6 months post operative the extraction socket in which the implant will be placed are class I&II

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients (American Society of Anesthesiologists I; ASA I).
* Age range (20-40) years.
* Good compliance with the plaque control instructions following initial therapy.
* Patients diagnosed with bone defect in the maxillary anterior esthetic zone (class 1 & 2)
* Availability for follow up and maintenance program.

Exclusion Criteria:

* Peri apically infected teeth
* Presence of smoking habit.
* Presence of occlusal interferences.
* Pregnant females.
* Vulnerable group of patients (handicapped, mentally retarded and prisoners) (according to the recommendation of esthetical committee of Faculty of Dentistry Ain Shams University).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
buccal bone thickness | at baseline and 9 months
  measuring the buccal bone thickness using CBCT

SECONDARY OUTCOMES:
soft tissue assessment using pink esthetic score | 9 months post opertive
  The pink esthetic score (PES) evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency, Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14
patient satisfaction | after 9 months
  questionnaire in which the scale is from (0 to 10) where 0 is completely unsatisfied and 10 totally satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abu el ela, Prof, Study Director — Faculty of dentistry ain shams university
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No